CLINICAL TRIAL: NCT04773470
Title: Implementation of Flexible Endoscopic Evaluation of Swallowing (FEES) and Standardized FEES Scores in the Diagnostic Work-up of Dysphagia in Spinal Muscular Atrophy - DYS-SMA Trial
Brief Title: Implementation of FEES in Spinal Muscle Atrophy
Acronym: DYS-SMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DYSSMA1
Record Dates: First submitted 2020-11-19; First posted 2021-02-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal Muscle Atrophy (Experimental): All patients with Spinal Muscle Atrophy type 1 to 4
  Interventions: Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing — Endoscopical swallowing study

SUMMARY:
The major aim of this project is to assess comprehensively frequency and extent of dysphagia and bulbar dysfunction in SMA1, 2, and 3 patients by applying FEES and validated dysphagia scores. Further aims are to follow changes of dysphagia over time in newly diagnosed patients, and in subjects starting treatment with one of the new therapeutic SMA drugs. Special attention will be paid to subjects treated with Risdiplam. If applicable, the data will be compared between groups receiving different drugs.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a progressive autosomal recessive neuromuscular disease characterized by premature degeneration of the 2nd motor neuron and a broad phenotype. SMA results from biallelic mutations in the SMN1 gene at 5q13. SMN1 encodes the SMN protein that is essential for proper function of the anterior horn cells. The estimated incidence is 1 per 6000-11 000 births. The classification of SMA is based on age at symptom onset and maximum motor function achieved. SMA1 patients develop symptoms within the first 6 months of life and do not achieve sitting without support. SMA2 patients typically show first symptoms from 6 to 18 months and never learn to walk. SMA3 patients display first clinical signs after the age of 18 months and achieve walking. Rarely, patients develop first symptoms in adulthood (SMA4). While defects in SMN1 are the cause of SMA, the severity of disease is related to the copy number of SMN2, a paralogous gene located next to SMN1 that differs from SMN1 by 5 nucleotides only. This results in a splicing defect reducing the amount of SMN protein produced by one copy of SMN2 to about 10%.

The clinical hallmarks of SMA are progressive muscle weakness and muscular atrophy. Scoliotic deformities, contractures, reduced head control, limited jaw closure, coughing difficulties, and impaired clearance of tracheal secretions are common problems. In many patients, bulbar muscle weakness including dysphagia represents a great diagnostic and therapeutic challenge.

Treatment of SMA remained purely symptomatic for many decades, but this has changed fundamentally within the last years, since several therapeutic agents have been developed targeting to correct causal disease mechanisms. Nusinersen, an antisense oligonucleotide modifying SMN2 splicing, has been approved in the US and in Europe. Onasemnogene abeparvovec, an AAV9-mediated gene therapy, provides patients with intact SMN1 copies and has also been licensed in the US and in Europe. Finally, Risdiplam, an oral splicing modifier acting on SMN2, has been approved in the US and is currently available in Germany for SMA1 and 2 patients via a compassionate use program. Data from two recent studies, FIREFISH (SMA1) and SUNFISH (SMA2/3) have shown significant improvements in motor and bulbar functions in Risdiplam treated individuals.

Although these new therapies will substantially modify the course of disease and improve the prognosis of SMA, the treatment of clinical symptoms and their diagnosis will remain challenging. Dysphagia of variable degree often necessitating artificial feeding to prevent malnutrition and low body weight occurs in all types of SMA. Poor sucking, swallowing difficulties, and inadequate mobilization of mucous with increased risk of aspiration and pneumonia are frequent in SMA1, while restricted jaw mobility and opening as well as weakness of the jaw muscles are common in SMA2 and 3. Altogether, dysphagia represents an important factor of morbidity in SMA, and adequate diagnosis and care of this symptom are essential to maintain quality of life. To achieve this, the application of validated diagnostic methods and scales are necessary. But until now, only a few retrospective studies with small numbers of patients or case reports dealing with dysphagia in SMA are on record, and no standardized assessments using validated tests have been applied. Moreover, no larger study has systematically analyzed which percentages of SMA1, 2, and 3 patients suffer from dysphagia, and no data are available about severity of dysphagia in the single types. Furthermore, it is not known, which effects on swallowing the new therapeutic agents have.

Flexible Endoscopic Evaluation of Swallowing (FEES) is the gold standard of swallowing imaging, but has not yet been comprehensively and prospectively used for analysis of the swallowing process in SMA. In patients with neurogenic dysphagia, validated dysphagia severity scores in tandem with FEES are used since many years, and allow early detection and improved management of swallowing disorders.

ELIGIBILITY:
Inclusion Criteria:

All patients with genetically determined 5q-linked SMA followed at the neuromuscular center Gießen

- Informed and written consent signed by the patient or a legal guardian

Exclusion Criteria:

* Physical illness that, according to its type and severity, could interfere with the planned assessments, could have an influence on the parameters to be investigated or could endanger the patient or test person during the course of the investigation.
* Pregnancy or lactation and a positive pregnancy test
* Acute suicidal tendency or external danger
* Poor general condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Secretion severity | Baseline
  Change in presence and severity of dysphagia examined via FEES and scored by Murray´s Secretions Severity Rating Scale Minimum value: 0 Maximum value: 3 Higher scores mean worse outcome
Dysphagia severity | Baseline
  Change in presence and severity of dysphagia examined via FEES and scored by Rosenbek´s Penetration-Aspiration-Scale Minimum value: 1 Maximum value: 8 Higher scores mean worse outcome
Pharyngeal residue severity | Baseline
  Change in presence and severity of dysphagia examined via FEES and scored by Yale Pharyngeal Residue Severity Rating Scale Minimum value: 1 Maximum value: 5 Higher scores mean worse outcome
Functional Oral Intake Scale | Baseline
  Assessment of functional oral intake over time. Scored via Functional Oral Intake Scale (FOIS-G, German version): Minimum value 1, maximum value 7; lower scores mean worse outcome
Severity of Dysphagia in Neuromuscular Diseases | Baseline
  Severity of dysphagia in neuromuscular diseases paired with necessity of oropharyngeal and endotracheal suction as measuered via Neuromuscular Disease Swallowing Status Scale; Minimum value 1, maximum value 8; lower scores mean worse outcome
Upper limb function | Baseline
  Assessment specifically designed for upper limb function in SMA patients: RULM-Test (Revised Upper Limb Module); minimum value 1, maximum value 37; lower values mean worse outcome
Functional motor abilites | Baseline
  Functional motor abilities as measured by HFSME-Test (Hammersmith Functional Motor Scale). Minimum value 0, maximum value 2; lower values mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Samra Hamzic, MA, Principal Investigator — University Giessen
Locations (1):
- University Hospital Giessen and Marburg, Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No